CLINICAL TRIAL: NCT03185598
Title: MACE and First Operating Room Systolic Blood Pressure in Patients Undergoing Non-cardiac Surgery Implications for the Hypertension Threshold
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, MD, Peking University First Hospital
Other Study IDs: ORSBPTHRE
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Major Adverse Cardiac-cerebral-kidney Event

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-MACE: no MACE occurred
- MACE: MACE occurred

SUMMARY:
To find the threshold of First operating room SBP above which MACE risk increases.

DETAILED DESCRIPTION:
To find the threshold of First operating room SBP above which MACE risk increases. By reviewing data from 2012-2017 in PKU first hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18-100yr non-cardiac surgery

Exclusion Criteria:

* missing data file

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 90342 eligible surgeries among 71164 unique patients included
Sampling Method: Non-Probability Sample
Enrollment: 90342 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days postoperatively
  major adverse cardiac-cerebral-kidney event

IPD SHARING:
Plan to Share IPD: No